CLINICAL TRIAL: NCT01676597
Title: Efficacy of Pentoxifylline and Rifaximin Combination in Pentoxifylline Refractory Clinical and Subclinical Hepatopulmonary Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-HPS-01
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Hepatopulmonary Syndrome
MeSH Terms: conditions — Hepatopulmonary Syndrome | interventions — Pentoxifylline; Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rifaximin and pentoxifylline (Experimental): Tab Rifaximin 400 mg thrice daily + Pentoxifylline 400 mg thrice daily for 12 weeks
  Interventions: Drug: Pentoxifylline and placebo
- pentoxifylline and placebo (Active Comparator): Tab Pentoxifylline 400 mg thrice daily + Placebo thrice daily for 12 weeks
  Interventions: Drug: pentoxifylline and rifaximin

INTERVENTIONS:
Drug: pentoxifylline and rifaximin — Tab Rifaximin 400 mg thrice daily + Pentoxifylline 400 mg thrice daily for 12 weeks
  Arms: pentoxifylline and placebo
Drug: Pentoxifylline and placebo — Tab Pentoxifylline 400 mg thrice daily + Placebo thrice daily for 12 weeks
  Arms: rifaximin and pentoxifylline

SUMMARY:
* The study will be a prospective open labelled double blinded randomized controlled study.
* The study will be conducted on patients admitted to Department of Hepatology from 2012 to 2014 at Institute of Liver and Biliary Sciences, New Delhi
* Patients diagnosed as having clinical or subclinical hepatopulmonary syndrome will be started on oral pentoxifylline therapy 400 mg thrice daily for 12 weeks.
* Patients not responding to this therapy will be given divided into 2 arms with one arm receiving additional Tab Rifaximin 400 mg thrice daily or placebo for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of portal hypertension (esophagogastric varices or portal hypertensive gastropathy identified on esophagogastroduodenoscopy, and/or varices seen on computerized tomography scan or ultrasound, and/or splenomegaly with no other explanation, and/or ascites with no other explanation)
2. Intrapulmonary vascular dilatations (IPVDs) diagnosed on contrast echocardiogram (CE)
3. AaDO2 > 15 mm Hg on standing room air arterial blood gas (ABG)
4. Ability and willingness to give informed consent

Exclusion Criteria:

* Age < 18 or > 64
* Intrinsic significant cardiopulmonary disease
* Inability to perform pulmonary function tests
* Moderate to severe Pulmonary hypertension
* Advanced hepatic encephalopathy
* Inadequate echocardiographic window to allow for accurate transthoracic contrast echocardiography
* Antibiotic use within the last one month
* Listed for liver transplant in next 4 weeks
* Current use of exogenous nitrates
* Active bacterial infections
* Known malignancy
* Known intolerance to Pentoxifylline or rifaximin

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Complete response after 3 months of treatment | 3 months

SECONDARY OUTCOMES:
Development of serious adverse effects leading to withdrawal of the drug | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Naveen Kumar, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India